CLINICAL TRIAL: NCT06611501
Title: Glycemic Regulation as Endometriosis Adjunct Treatment
Acronym: GREAT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Jessica Shim, Assistant Professor, Division of Gynecology, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-P00049391
Record Dates: First submitted 2024-09-10; First posted 2024-09-25 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Pelvic Pain; Endometriosis
Keywords: Pelvic pain; Pain; Metformin; Chronic pain; Physiological Effects of Drugs; Endometriosis; Female Urogenital Diseases; Genital Diseases, Female
MeSH Terms: conditions — Pelvic Pain; Endometriosis; Pain; Chronic Pain; Female Urogenital Diseases; Genital Diseases, Female | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo tablets orally daily for a total of 6 months of treatment.
  Interventions: Drug: Placebo
- Metformin (Experimental): metformin hydrochloride 500 mg capsules daily for a total of 6 months of treatment
  Interventions: Drug: Metformin Hydrochloride

INTERVENTIONS:
Drug: Metformin Hydrochloride — Metformin dosage titrated from 500 mg/daily for 2 weeks, then 1000 mg/daily for 2 weeks, 1500 mg/daily for 2 weeks, and then achieving 2000 mg/daily for a duration of 6 months of treatment.
  Arms: Metformin
Drug: Placebo — 1 tablet orally with evening meal for 2 weeks, then 1 tablet twice daily for 2 weeks, then 3 tablets split twice daily for 2 weeks, then 4 tablets split twice daily, for a total of 6 months of treatment.
  Other Names: Placebo capsule
  Arms: Placebo

SUMMARY:
The goal of this pilot trial is to learn if a novel non-hormonal treatment, metformin hydrochloride, works to treat pelvic pain in young women with endometriosis. The main questions it aims to answer are:

* Is metformin superior to placebo in alleviating pain symptoms in young women with endometriosis?
* Does metformin alter systemic inflammatory markers over 6 months in young women with endometriosis?

Researchers will compare metformin to a placebo (a look-alike substance that contains no drug) to see if metformin works to treat pelvic pain.

Participants will:

* Take drug metformin or a placebo every day for 6 months
* Visit the clinic three times: once at baseline (pre-treatment), once at 3 months, and once at 6 months
* Keep a daily symptom diary to track pain, bleeding, and usage of any pain medications

DETAILED DESCRIPTION:
Endometriosis is a chronic illness defined by the presence of endometrial glands and stroma outside the uterine lining. While prevalence estimates vary depending on the population studied, endometriosis is thought to affect approximately one in ten reproductive aged women, up to 50% of women with infertility, and up to 70% of adolescents with chronic pelvic pain. Over 10 million women in the United States have endometriosis and incur significantly higher direct and indirect healthcare costs than those without. Annual health care costs are estimated at $100 billion in the United States alone. While the majority of patients report the onset of endometriosis symptoms during adolescence, delays in diagnosis are common and range from 7 to 12 years. During these delays, women may suffer from debilitating symptoms interfering with school and social activities, and commonly experience reduced health-related quality of life and work productivity. When left untreated, endometriosis can progress significantly in over 50% of patients and result in a higher stage of disease. Therefore, timely intervention and maintenance of therapy is critical for preventing the progression of disease and patient burden.

Therapeutic options for endometriosis include surgical and medical management. Because surgery is not curative, long-term medical therapy is often advised to prevent recurrence of symptoms and retard the progression of disease. Nonsteroidal anti-inflammatory drugs (NSAIDs) are commonly used for endometriosis-related pain but do not remove or decrease deposits of ectopic endometrium. Hormonal therapies are the mainstay of medical therapy as they can inhibit prostaglandin production that contributes to pain, and cause decidualization and atrophy of ectopic endometrial tissue. Unfortunately, hormonal treatments have varied degrees of success and no data support one treatment over another. Additionally, the treatment choice may be limited to medication side effects, availability, costs, and contraceptive needs. Hormonal treatments do not cure endometriosis; 11-19% of women may not experience any relief with medical therapy, and up to a third of women experience recurrence of pain symptoms after treatment cessation. Additionally, as endometriosis is predominantly a disease of young reproductive-aged women, patients may desire a treatment with a different mechanism of action that does not impact ovarian function and fertility. There remains an unmet clinical need among women with endometriosis for effective and well-tolerated medical therapies.

Metformin, an insulin-sensitizing oral biguanide, is approved for the treatment of type 2 diabetes. Several published studies using in vitro and animal models have implicated metformin with a regression of endometriotic implants and reduction of inflammatory activity. Yet, the mechanisms of action of metformin remain to be further elucidated. Only one prospective study to date has investigated the use of metformin in humans as monotherapy for endometriosis; this study had substantial limitations. Further investigation will be improved with participant and provider blinding, use of validated pain measures, and inclusion of a broader population of patients affected by endometriosis. A randomized clinical trial is necessary to investigate the mechanisms and efficacy of metformin as an anti-endometriotic drug.

ELIGIBILITY:
Inclusion Criteria:

* Female with surgically confirmed endometriosis, determined at laparoscopy
* Current use for at least 2 months duration of a consistent hormonal therapy for endometriosis (either combination hormonal contraceptives or progestin-only therapy)
* Current pelvic pain (score ≥ 3 on Visual Analog Scale) that has been present for at least 2 months prior to enrollment
* Age 15 years to 35 years and premenopausal
* Willingness to comply with visit schedule and protocol

Exclusion Criteria:

* Pre-menarche or post-menopause
* Diagnosis of Type 1 or Type 2 Diabetes Mellitus
* Severe renal dysfunction (creatinine >1.4 mg/dL or eGFR below 45 mL/minute/1.73 m2
* History of lactic acidosis or diabetic ketoacidosis
* ALT or AST > 2.5 times the upper limit of normal
* Significant mental or chronic systemic illness that might confound pain assessment or the inability to complete the study
* Current/planning pregnancy or breastfeeding
* Inability to read English

Ages: 15 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain assessed by the Brief Pain Inventory Interference Scale (BPI) over 6 months | once at each of the three visits (at baseline, 3 months, 6 months)
  The BPI Interference Scale is a 7-item composite pain measurement. This self-report measure assesses the extent to which pain interferes with various components of physical and emotional functioning and sleep. The items in this scale can be grouped into those that assess physical functioning (general activity; walking ability; normal work, including both work outside the home and housework), those that assess emotional functioning (mood; relations with people; enjoyment of life), and a single item that assess the extent to which pain interferes with sleep. The arithmetic mean of the seven interference items can be used as a measure of pain interference. The BPI is anchored between a scale of zero (no pain/interference) to ten (maximum pain/interference). The magnitude of treatment-associated change in BPI Interference Scale scores in open-label and randomized clinical trials ranges from 1 to 3 points, depending on the specific pain conditions and treatments studied.
Change in pain severity measured by Visual Analog Scale (VAS) over 6 months | once at each of the three visits (at baseline, 3 months, 6 months)
  VAS: A measurement of pain intensity, assessed by a 0 to 10 numerical rating scale, to rate maximum and average pain intensity over the preceding 7 days. Higher scores indicate more severe pain intensity.
Change in emotional functioning assessed by Beck Depression Inventory-II (BDI) over 6 months | once at each of the three visits (at baseline, 3 months, 6 months)
  The BDI is a 21-item self-report instrument that provides a rapid assessment of depressive symptoms. BDI has been used in many studies of chronic pain, including chronic pelvic pain and endometriosis. Total scores on the BDI range from 0 to 63. The BDI takes about 5-10 minutes to complete. Scores below 13 should be considered to reflect "minimal or no" depression, with score ranges of 14 to 19, 20 to 28, and 29 to 63 reflect "mild to moderate," "moderate to severe," and "severe" depression, respectively.
Change in ratings of overall improvement assessed by the Patient Global Impression of Change scale (PGIC) | once at each of the three visits (at baseline, 3 months, 6 months)
  The PGIC is a seven-point single-item scale with options ranging from 'very much worse' to 'very much improved'. There has been widespread use of the PGIC in recent endometriosis clinical trials, as it readily interprets a person's evaluation of the importance of their improvement or worsening.

SECONDARY OUTCOMES:
Change in quality of life, measured via Endometriosis Health Profile-30 (EHP-30) | once at each of the three visits (at baseline, 3 months, 6 months)
  The EHP-30 is a reliable instrument and recommended by the American Society for Reproductive Medicine and the European Society for Human Reproduction and Embryology. The questionnaire includes 30 questions in five subcategories, with each category addressing specific problem areas of pain, control and powerlessness, emotional wellbeing, social support, and self-image.
Changes in sexual satisfaction for participants who are sexually active measured by the New Sexual Satisfaction Scale | once at each of the three visits (at baseline, 3 months, 6 months)
  The NSSS is a 20-item measure assessing sexual sensations, sexual presence/awareness, sexual exchange, emotional connection/closeness, and sexual activity. The full scale takes 5 minutes to complete.
Complete health and medication history assessed by the World Endometriosis Research Foundation (WERF) questionnaire | once at each of the three visits (at baseline, 3 months, 6 months)
  Study participants will complete an expanded version of the WERF questionnaire for a complete health and medication history
Changes in serum angiogenic/inflammatory markers | once at each of the three visits (at baseline, 3 months, 6 months)
  Serum samples will also be obtained for measures of inflammation, to test the hypothesis that endometriosis-relevant inflammatory markers will decrease over time in patients treated with metformin compared to those receiving placebo. These markers will include IL-6, IL-8, and VEGF based on the results of prior studies in which metformin appeared to reduce these levels in humans with endometriosis and from endometriotic implants in rats. C-reactive protein (CRP) will also be assessed; CRP has been shown to be upregulated, especially when examined with a high sensitivity assay making it possible to detect subclinical inflammation in women with endometriosis.

OTHER OUTCOMES:
Changes in school and/or work attendance | once at each of the three visits (at baseline, 3 months, 6 months)
  School and/or work attendance will be assessed at each visit.
Change in pregnancy status | once at each of the three visits (at baseline, 3 months, 6 months)
  Urine pregnancy test throughout the study as current pregnancy is an exclusion criteria
Changes in serum lactate levels | baseline, three and six months if needed
  Serum lactate will be measured at baseline and then possibly at three and six months, if needed.
Changes in pain | daily for 6 months
  Subjects will keep a daily symptom diary to track pain for 6 months.
Incidence of vaginal bleeding over six months | daily for 6 months
  Measurement of the incidence of vaginal bleeding using a daily symptom diary to document the presence/absence of vaginal bleeding
Usage of any pain medications (both prescription and over the counter) | daily for 6 months
  Usage of any pain medications (both prescription and over the counter) tracked in a daily symptom diary for 6 months
Changes in height | once at each of the three visits (at baseline, 3 months, 6 months)
  Height, in cm, will be obtained at each study visit (at baseline, 3 months, and 6 months).
Changes in weight | once at each of the three visits (at baseline, 3 months, 6 months)
  Study subjects will have their weight obtained at each study visit given the potential impact on weight by metformin.
Changes in serum insulin c-peptide level | at baseline and 6 months
  Serum insulin c-peptide levels will be collected at baseline and again at 6-months given metformin impact on lowering c-peptide levels.
Changes in hemoglobin and mean corpuscular volume | at baseline and 6 months
  A Complete Blood Count (CBC) will be collected at baseline and again at 6-months due to the potential adverse effect of megaloblastic anemia by metformin, which would be detected by the hemoglobin and mean corpuscular volume.
Changes in vitamin B12 levels | at baseline and 6 months
  Serum vitamin B12 levels will be obtained at baseline and at 6 months due to the possible adverse effect of vitamin b12 deficiency by metformin
Changes in lipid levels | at baseline and 6 months
  A lipid panel will be collected at baseline and again at 6-months due to the potential lipid-lowering activity of metformin.
Changes in hemoglobin A1c | once at each of the three visits (at baseline, 3 months, 6 months)
  At each study visit, (baseline, 3 months, and 6 months), HbA1c will be assessed serially given the glycemic impact and effect of reducing HbA1c by metformin.
Changes in metabolic panel | once at each of the three visits (at baseline, 3 months, 6 months)
  At each study visit, (baseline, 3 months, and 6 months), a comprehensive metabolic panel will be assessed serially to monitor for any potential kidney impairment that might affect continuation of treatment or changes in electrolytes in the setting of gastrointestinal distress.
Changes in temperature | once at each of the three visits (at baseline, 3 months, 6 months)
  A physical exam will be conducted at baseline, three months, and six months to obtain changes in temperature.
Changes in heart rate | once at each of the three visits (at baseline, 3 months, 6 months)
  A physical exam will be conducted at baseline, three months, and six months to obtain changes in heart rate.
Changes in blood pressure | once at each of the three visits (at baseline, 3 months, 6 months)
  A physical exam will be conducted at baseline, three months, and six months to obtain changes in blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Shim, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared so that patient privacy and confidentiality is maintained during this study.

REFERENCES:
- [Background] Laufer MR, Goitein L, Bush M, Cramer DW, Emans SJ. Prevalence of endometriosis in adolescent girls with chronic pelvic pain not responding to conventional therapy. J Pediatr Adolesc Gynecol. 1997 Nov;10(4):199-202. doi: 10.1016/s1083-3188(97)70085-8. PMID 9391902
- [Background] Nnoaham KE, Hummelshoj L, Webster P, d'Hooghe T, de Cicco Nardone F, de Cicco Nardone C, Jenkinson C, Kennedy SH, Zondervan KT; World Endometriosis Research Foundation Global Study of Women's Health consortium. Impact of endometriosis on quality of life and work productivity: a multicenter study across ten countries. Fertil Steril. 2011 Aug;96(2):366-373.e8. doi: 10.1016/j.fertnstert.2011.05.090. Epub 2011 Jun 30. PMID 21718982
- [Background] Brown J, Crawford TJ, Allen C, Hopewell S, Prentice A. Nonsteroidal anti-inflammatory drugs for pain in women with endometriosis. Cochrane Database Syst Rev. 2017 Jan 23;1(1):CD004753. doi: 10.1002/14651858.CD004753.pub4. PMID 28114727
- [Background] Suda K, Nakaoka H, Yoshihara K, Ishiguro T, Tamura R, Mori Y, Yamawaki K, Adachi S, Takahashi T, Kase H, Tanaka K, Yamamoto T, Motoyama T, Inoue I, Enomoto T. Clonal Expansion and Diversification of Cancer-Associated Mutations in Endometriosis and Normal Endometrium. Cell Rep. 2018 Aug 14;24(7):1777-1789. doi: 10.1016/j.celrep.2018.07.037. PMID 30110635
- [Background] Becker CM, Bokor A, Heikinheimo O, Horne A, Jansen F, Kiesel L, King K, Kvaskoff M, Nap A, Petersen K, Saridogan E, Tomassetti C, van Hanegem N, Vulliemoz N, Vermeulen N; ESHRE Endometriosis Guideline Group. ESHRE guideline: endometriosis. Hum Reprod Open. 2022 Feb 26;2022(2):hoac009. doi: 10.1093/hropen/hoac009. eCollection 2022. PMID 35350465
- [Background] Hossain MM, Nakayama K, Shanta K, Razia S, Ishikawa M, Ishibashi T, Yamashita H, Sato S, Iida K, Kanno K, Ishikawa N, Kiyono T, Kyo S. Establishment of a Novel In Vitro Model of Endometriosis with Oncogenic KRAS and PIK3CA Mutations for Understanding the Underlying Biology and Molecular Pathogenesis. Cancers (Basel). 2021 Jun 25;13(13):3174. doi: 10.3390/cancers13133174. PMID 34202354
- [Background] Hopkins BD, Pauli C, Du X, Wang DG, Li X, Wu D, Amadiume SC, Goncalves MD, Hodakoski C, Lundquist MR, Bareja R, Ma Y, Harris EM, Sboner A, Beltran H, Rubin MA, Mukherjee S, Cantley LC. Suppression of insulin feedback enhances the efficacy of PI3K inhibitors. Nature. 2018 Aug;560(7719):499-503. doi: 10.1038/s41586-018-0343-4. Epub 2018 Jul 4. PMID 30051890
- [Background] Qiang P, Shao Y, Sun YP, Zhang J, Chen LJ. Metformin inhibits proliferation and migration of endometrial cancer cells through regulating PI3K/AKT/MDM2 pathway. Eur Rev Med Pharmacol Sci. 2019 Feb;23(4):1778-1785. doi: 10.26355/eurrev_201902_17140. PMID 30840303
- [Background] Shu Y, Sheardown SA, Brown C, Owen RP, Zhang S, Castro RA, Ianculescu AG, Yue L, Lo JC, Burchard EG, Brett CM, Giacomini KM. Effect of genetic variation in the organic cation transporter 1 (OCT1) on metformin action. J Clin Invest. 2007 May;117(5):1422-31. doi: 10.1172/JCI30558. PMID 17476361
- [Background] Oner G, Ozcelik B, Ozgun MT, Serin IS, Ozturk F, Basbug M. The effects of metformin and letrozole on endometriosis and comparison of the two treatment agents in a rat model. Hum Reprod. 2010 Apr;25(4):932-7. doi: 10.1093/humrep/deq016. Epub 2010 Feb 3. PMID 20133323
- [Background] Yilmaz B, Sucak A, Kilic S, Aksakal O, Aksoy Y, Lortlar N, Sut N, Gungor T. Metformin regresses endometriotic implants in rats by improving implant levels of superoxide dismutase, vascular endothelial growth factor, tissue inhibitor of metalloproteinase-2, and matrix metalloproteinase-9. Am J Obstet Gynecol. 2010 Apr;202(4):368.e1-8. doi: 10.1016/j.ajog.2009.10.873. Epub 2009 Dec 29. PMID 20035912
- [Background] Zhang H, Xue J, Li M, Zhao X, Wei D, Li C. Metformin regulates stromal-epithelial cells communication via Wnt2/beta-catenin signaling in endometriosis. Mol Cell Endocrinol. 2015 Sep 15;413:61-5. doi: 10.1016/j.mce.2015.06.011. Epub 2015 Jun 24. PMID 26116230
- [Background] Davies MJ, D'Alessio DA, Fradkin J, Kernan WN, Mathieu C, Mingrone G, Rossing P, Tsapas A, Wexler DJ, Buse JB. Management of Hyperglycemia in Type 2 Diabetes, 2018. A Consensus Report by the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD). Diabetes Care. 2018 Dec;41(12):2669-2701. doi: 10.2337/dci18-0033. Epub 2018 Oct 4. PMID 30291106
- [Background] Rowan JA, Hague WM, Gao W, Battin MR, Moore MP; MiG Trial Investigators. Metformin versus insulin for the treatment of gestational diabetes. N Engl J Med. 2008 May 8;358(19):2003-15. doi: 10.1056/NEJMoa0707193. PMID 18463376
- [Background] Velazquez EM, Mendoza S, Hamer T, Sosa F, Glueck CJ. Metformin therapy in polycystic ovary syndrome reduces hyperinsulinemia, insulin resistance, hyperandrogenemia, and systolic blood pressure, while facilitating normal menses and pregnancy. Metabolism. 1994 May;43(5):647-54. doi: 10.1016/0026-0495(94)90209-7. PMID 8177055
- [Background] Jackson RA, Hawa MI, Jaspan JB, Sim BM, Disilvio L, Featherbe D, Kurtz AB. Mechanism of metformin action in non-insulin-dependent diabetes. Diabetes. 1987 May;36(5):632-40. doi: 10.2337/diab.36.5.632. PMID 3552795
- [Background] Wu H, Esteve E, Tremaroli V, Khan MT, Caesar R, Manneras-Holm L, Stahlman M, Olsson LM, Serino M, Planas-Felix M, Xifra G, Mercader JM, Torrents D, Burcelin R, Ricart W, Perkins R, Fernandez-Real JM, Backhed F. Metformin alters the gut microbiome of individuals with treatment-naive type 2 diabetes, contributing to the therapeutic effects of the drug. Nat Med. 2017 Jul;23(7):850-858. doi: 10.1038/nm.4345. Epub 2017 May 22. PMID 28530702
- [Background] Palmer SC, Mavridis D, Nicolucci A, Johnson DW, Tonelli M, Craig JC, Maggo J, Gray V, De Berardis G, Ruospo M, Natale P, Saglimbene V, Badve SV, Cho Y, Nadeau-Fredette AC, Burke M, Faruque L, Lloyd A, Ahmad N, Liu Y, Tiv S, Wiebe N, Strippoli GF. Comparison of Clinical Outcomes and Adverse Events Associated With Glucose-Lowering Drugs in Patients With Type 2 Diabetes: A Meta-analysis. JAMA. 2016 Jul 19;316(3):313-24. doi: 10.1001/jama.2016.9400. PMID 27434443
- [Background] Takemura Y, Osuga Y, Yoshino O, Hasegawa A, Hirata T, Hirota Y, Nose E, Morimoto C, Harada M, Koga K, Tajima T, Yano T, Taketani Y. Metformin suppresses interleukin (IL)-1beta-induced IL-8 production, aromatase activation, and proliferation of endometriotic stromal cells. J Clin Endocrinol Metab. 2007 Aug;92(8):3213-8. doi: 10.1210/jc.2006-2486. Epub 2007 May 15. PMID 17504902
- [Background] Nodler JL, DiVasta AD, Vitonis AF, Karevicius S, Malsch M, Sarda V, Fadayomi A, Harris HR, Missmer SA. Supplementation with vitamin D or omega-3 fatty acids in adolescent girls and young women with endometriosis (SAGE): a double-blind, randomized, placebo-controlled trial. Am J Clin Nutr. 2020 Jul 1;112(1):229-236. doi: 10.1093/ajcn/nqaa096. PMID 32453393
- [Background] DiVasta AD, Stamoulis C, Gallagher JS, Laufer MR, Anchan R, Hornstein MD. Nonhormonal therapy for endometriosis: a randomized, placebo-controlled, pilot study of cabergoline versus norethindrone acetate. F S Rep. 2021 Jul 24;2(4):454-461. doi: 10.1016/j.xfre.2021.07.003. eCollection 2021 Dec. PMID 34934987
- [Background] Yanovski JA, Krakoff J, Salaita CG, McDuffie JR, Kozlosky M, Sebring NG, Reynolds JC, Brady SM, Calis KA. Effects of metformin on body weight and body composition in obese insulin-resistant children: a randomized clinical trial. Diabetes. 2011 Feb;60(2):477-85. doi: 10.2337/db10-1185. Epub 2011 Jan 12. PMID 21228310
- [Background] Adeyemo MA, McDuffie JR, Kozlosky M, Krakoff J, Calis KA, Brady SM, Yanovski JA. Effects of metformin on energy intake and satiety in obese children. Diabetes Obes Metab. 2015 Apr;17(4):363-70. doi: 10.1111/dom.12426. Epub 2015 Jan 11. PMID 25483291
- [Background] Srinivasan S, Ambler GR, Baur LA, Garnett SP, Tepsa M, Yap F, Ward GM, Cowell CT. Randomized, controlled trial of metformin for obesity and insulin resistance in children and adolescents: improvement in body composition and fasting insulin. J Clin Endocrinol Metab. 2006 Jun;91(6):2074-80. doi: 10.1210/jc.2006-0241. Epub 2006 Apr 4. PMID 16595599
- [Background] Mauras N, DelGiorno C, Hossain J, Bird K, Killen K, Merinbaum D, Weltman A, Damaso L, Balagopal P. Metformin use in children with obesity and normal glucose tolerance--effects on cardiovascular markers and intrahepatic fat. J Pediatr Endocrinol Metab. 2012;25(1-2):33-40. doi: 10.1515/jpem-2011-0450. PMID 22570948
- [Background] Dworkin RH, Turk DC, Wyrwich KW, Beaton D, Cleeland CS, Farrar JT, Haythornthwaite JA, Jensen MP, Kerns RD, Ader DN, Brandenburg N, Burke LB, Cella D, Chandler J, Cowan P, Dimitrova R, Dionne R, Hertz S, Jadad AR, Katz NP, Kehlet H, Kramer LD, Manning DC, McCormick C, McDermott MP, McQuay HJ, Patel S, Porter L, Quessy S, Rappaport BA, Rauschkolb C, Revicki DA, Rothman M, Schmader KE, Stacey BR, Stauffer JW, von Stein T, White RE, Witter J, Zavisic S. Interpreting the clinical importance of treatment outcomes in chronic pain clinical trials: IMMPACT recommendations. J Pain. 2008 Feb;9(2):105-21. doi: 10.1016/j.jpain.2007.09.005. Epub 2007 Dec 11. PMID 18055266
- [Background] Keller S, Bann CM, Dodd SL, Schein J, Mendoza TR, Cleeland CS. Validity of the brief pain inventory for use in documenting the outcomes of patients with noncancer pain. Clin J Pain. 2004 Sep-Oct;20(5):309-18. doi: 10.1097/00002508-200409000-00005. PMID 15322437
- [Background] Smarr KL, Keefer AL. Measures of depression and depressive symptoms: Beck Depression Inventory-II (BDI-II), Center for Epidemiologic Studies Depression Scale (CES-D), Geriatric Depression Scale (GDS), Hospital Anxiety and Depression Scale (HADS), and Patient Health Questionnaire-9 (PHQ-9). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S454-66. doi: 10.1002/acr.20556. No abstract available. PMID 22588766
- [Background] Pokrzywinski R, Soliman AM, Surrey E, Snabes MC, Coyne KS. Psychometric assessment of the PROMIS Fatigue Short Form 6a in women with moderate-to-severe endometriosis-associated pain. J Patient Rep Outcomes. 2020 Oct 27;4(1):86. doi: 10.1186/s41687-020-00257-y. PMID 33108543
- [Background] Bourdel N, Chauvet P, Billone V, Douridas G, Fauconnier A, Gerbaud L, Canis M. Systematic review of quality of life measures in patients with endometriosis. PLoS One. 2019 Jan 10;14(1):e0208464. doi: 10.1371/journal.pone.0208464. eCollection 2019. PMID 30629598
- [Background] Vitonis AF, Vincent K, Rahmioglu N, Fassbender A, Buck Louis GM, Hummelshoj L, Giudice LC, Stratton P, Adamson GD, Becker CM, Zondervan KT, Missmer SA; WERF EPHect Working Group. World Endometriosis Research Foundation Endometriosis Phenome and Biobanking Harmonization Project: II. Clinical and covariate phenotype data collection in endometriosis research. Fertil Steril. 2014 Nov;102(5):1223-32. doi: 10.1016/j.fertnstert.2014.07.1244. Epub 2014 Sep 22. PMID 25256930
- [Background] Othman Eel-D, Hornung D, Salem HT, Khalifa EA, El-Metwally TH, Al-Hendy A. Serum cytokines as biomarkers for nonsurgical prediction of endometriosis. Eur J Obstet Gynecol Reprod Biol. 2008 Apr;137(2):240-6. doi: 10.1016/j.ejogrb.2007.05.001. Epub 2007 Jun 19. PMID 17582674
- [Background] Bedaiwy MA, Falcone T, Sharma RK, Goldberg JM, Attaran M, Nelson DR, Agarwal A. Prediction of endometriosis with serum and peritoneal fluid markers: a prospective controlled trial. Hum Reprod. 2002 Feb;17(2):426-31. doi: 10.1093/humrep/17.2.426. PMID 11821289
- [Background] Xavier P, Belo L, Beires J, Rebelo I, Martinez-de-Oliveira J, Lunet N, Barros H. Serum levels of VEGF and TNF-alpha and their association with C-reactive protein in patients with endometriosis. Arch Gynecol Obstet. 2006 Jan;273(4):227-31. doi: 10.1007/s00404-005-0080-4. Epub 2005 Oct 6. PMID 16208475
- [Background] Karbalaee-Hasani A, Khadive T, Eskandari M, Shahidi S, Mosavi M, Nejadebrahimi Z, Khalkhali L, Sangdari A, Mohammadi D, Soltani A, Khodabandehloo H, Hosseini H, Koushki M. Effect of Metformin on Circulating Levels of Inflammatory Markers in Patients With Type 2 Diabetes: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Ann Pharmacother. 2021 Sep;55(9):1096-1109. doi: 10.1177/1060028020985303. Epub 2021 Jan 7. PMID 33412927
- [Background] Seifarth C, Schehler B, Schneider HJ. Effectiveness of metformin on weight loss in non-diabetic individuals with obesity. Exp Clin Endocrinol Diabetes. 2013 Jan;121(1):27-31. doi: 10.1055/s-0032-1327734. Epub 2012 Nov 12. PMID 23147210
- [Background] Kujawska-Luczak M, Musialik K, Szulinska M, Swora-Cwynar E, Kargulewicz A, Grzymislawska M, Pupek-Musialik D, Bogdanski P. The effect of orlistat versus metformin on body composition and insulin resistance in obese premenopausal women: 3-month randomized prospective open-label study. Arch Med Sci. 2017 Jun;13(4):725-731. doi: 10.5114/aoms.2016.62014. Epub 2016 Aug 29. PMID 28721138
- [Background] DeFronzo RA, Goodman AM. Efficacy of metformin in patients with non-insulin-dependent diabetes mellitus. The Multicenter Metformin Study Group. N Engl J Med. 1995 Aug 31;333(9):541-9. doi: 10.1056/NEJM199508313330902. PMID 7623902
- [Background] Reese KA, Reddy S, Rock JA. Endometriosis in an adolescent population: the Emory experience. J Pediatr Adolesc Gynecol. 1996 Aug;9(3):125-8. doi: 10.1016/s1083-3188(96)70021-9. PMID 8795787
- [Background] Fujita Y, Inagaki N. Metformin: New Preparations and Nonglycemic Benefits. Curr Diab Rep. 2017 Jan;17(1):5. doi: 10.1007/s11892-017-0829-8. PMID 28116648
- [Background] Kashi Z, Mahrooz A, Kianmehr A, Alizadeh A. The Role of Metformin Response in Lipid Metabolism in Patients with Recent-Onset Type 2 Diabetes: HbA1c Level as a Criterion for Designating Patients as Responders or Nonresponders to Metformin. PLoS One. 2016 Mar 15;11(3):e0151543. doi: 10.1371/journal.pone.0151543. eCollection 2016. PMID 26978661
- [Background] Abrao MS, Podgaec S, Filho BM, Ramos LO, Pinotti JA, de Oliveira RM. The use of biochemical markers in the diagnosis of pelvic endometriosis. Hum Reprod. 1997 Nov;12(11):2523-7. doi: 10.1093/humrep/12.11.2523. PMID 9436699
- [Background] May KE, Conduit-Hulbert SA, Villar J, Kirtley S, Kennedy SH, Becker CM. Peripheral biomarkers of endometriosis: a systematic review. Hum Reprod Update. 2010 Nov-Dec;16(6):651-74. doi: 10.1093/humupd/dmq009. Epub 2010 May 12. PMID 20462942
- [Background] Pizzo A, Salmeri FM, Ardita FV, Sofo V, Tripepi M, Marsico S. Behaviour of cytokine levels in serum and peritoneal fluid of women with endometriosis. Gynecol Obstet Invest. 2002;54(2):82-7. doi: 10.1159/000067717. PMID 12566749
- [Background] Ohata Y, Harada T, Miyakoda H, Taniguchi F, Iwabe T, Terakawa N. Serum interleukin-8 levels are elevated in patients with ovarian endometrioma. Fertil Steril. 2008 Oct;90(4):994-9. doi: 10.1016/j.fertnstert.2007.07.1355. Epub 2008 Jul 16. PMID 18635170
- [Background] Pellicer A, Albert C, Mercader A, Bonilla-Musoles F, Remohi J, Simon C. The follicular and endocrine environment in women with endometriosis: local and systemic cytokine production. Fertil Steril. 1998 Sep;70(3):425-31. doi: 10.1016/s0015-0282(98)00204-0. PMID 9757870
- [Background] Stulhofer A, Busko V, Brouillard P. Development and bicultural validation of the new sexual satisfaction scale. J Sex Res. 2010 Jul;47(4):257-68. doi: 10.1080/00224490903100561. PMID 19629836
- [Background] van de Burgt TJ, Hendriks JC, Kluivers KB. Quality of life in endometriosis: evaluation of the Dutch-version Endometriosis Health Profile-30 (EHP-30). Fertil Steril. 2011 Apr;95(5):1863-5. doi: 10.1016/j.fertnstert.2010.11.009. Epub 2010 Dec 3. PMID 21122838
- [Background] Jones G, Kennedy S, Barnard A, Wong J, Jenkinson C. Development of an endometriosis quality-of-life instrument: The Endometriosis Health Profile-30. Obstet Gynecol. 2001 Aug;98(2):258-64. doi: 10.1016/s0029-7844(01)01433-8. PMID 11506842
- [Background] Waller KG, Shaw RW. Endometriosis, pelvic pain, and psychological functioning. Fertil Steril. 1995 Apr;63(4):796-800. doi: 10.1016/s0015-0282(16)57484-6. PMID 7890065
- [Background] Kames LD, Rapkin AJ, Naliboff BD, Afifi S, Ferrer-Brechner T. Effectiveness of an interdisciplinary pain management program for the treatment of chronic pelvic pain. Pain. 1990 Apr;41(1):41-46. doi: 10.1016/0304-3959(90)91107-T. PMID 2352765
- [Background] Vincent K, Kennedy S, Stratton P. Pain scoring in endometriosis: entry criteria and outcome measures for clinical trials. Report from the Art and Science of Endometriosis meeting. Fertil Steril. 2010 Jan;93(1):62-7. doi: 10.1016/j.fertnstert.2008.09.056. Epub 2008 Nov 5. PMID 18990378
- [Background] Raichle KA, Osborne TL, Jensen MP, Cardenas D. The reliability and validity of pain interference measures in persons with spinal cord injury. J Pain. 2006 Mar;7(3):179-86. doi: 10.1016/j.jpain.2005.10.007. PMID 16516823
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Bourdel N, Alves J, Pickering G, Ramilo I, Roman H, Canis M. Systematic review of endometriosis pain assessment: how to choose a scale? Hum Reprod Update. 2015 Jan-Feb;21(1):136-52. doi: 10.1093/humupd/dmu046. Epub 2014 Sep 1. PMID 25180023
- [Background] Siavash M, Tabbakhian M, Sabzghabaee AM, Razavi N. Severity of Gastrointestinal Side Effects of Metformin Tablet Compared to Metformin Capsule in Type 2 Diabetes Mellitus Patients. J Res Pharm Pract. 2017 Apr-Jun;6(2):73-76. doi: 10.4103/jrpp.JRPP_17_2. PMID 28616428
- [Background] Rojas LB, Gomes MB. Metformin: an old but still the best treatment for type 2 diabetes. Diabetol Metab Syndr. 2013 Feb 15;5(1):6. doi: 10.1186/1758-5996-5-6. PMID 23415113
- [Background] Reiser E, Lanbach J, Bottcher B, Toth B. Non-Hormonal Treatment Options for Regulation of Menstrual Cycle in Adolescents with PCOS. J Clin Med. 2022 Dec 21;12(1):67. doi: 10.3390/jcm12010067. PMID 36614868
- [Background] Flyckt R, Kim S, Falcone T. Surgical Management of Endometriosis in Patients with Chronic Pelvic Pain. Semin Reprod Med. 2017 Jan;35(1):54-64. doi: 10.1055/s-0036-1597306. Epub 2017 Jan 3. PMID 28049215
- [Background] Maruthur NM, Tseng E, Hutfless S, Wilson LM, Suarez-Cuervo C, Berger Z, Chu Y, Iyoha E, Segal JB, Bolen S. Diabetes Medications as Monotherapy or Metformin-Based Combination Therapy for Type 2 Diabetes: A Systematic Review and Meta-analysis. Ann Intern Med. 2016 Jun 7;164(11):740-51. doi: 10.7326/M15-2650. Epub 2016 Apr 19. PMID 27088241
- [Background] Stumvoll M, Nurjhan N, Perriello G, Dailey G, Gerich JE. Metabolic effects of metformin in non-insulin-dependent diabetes mellitus. N Engl J Med. 1995 Aug 31;333(9):550-4. doi: 10.1056/NEJM199508313330903. PMID 7623903
- [Background] LaMoia TE, Shulman GI. Cellular and Molecular Mechanisms of Metformin Action. Endocr Rev. 2021 Jan 28;42(1):77-96. doi: 10.1210/endrev/bnaa023. PMID 32897388
- [Background] Rena G, Hardie DG, Pearson ER. The mechanisms of action of metformin. Diabetologia. 2017 Sep;60(9):1577-1585. doi: 10.1007/s00125-017-4342-z. Epub 2017 Aug 3. PMID 28776086
- [Background] Tang T, Glanville J, Orsi N, Barth JH, Balen AH. The use of metformin for women with PCOS undergoing IVF treatment. Hum Reprod. 2006 Jun;21(6):1416-25. doi: 10.1093/humrep/del025. Epub 2006 Feb 24. PMID 16501038
- [Background] Khattab S, Fotouh IA, Mohesn IA, Metwally M, Moaz M. Use of metformin for prevention of ovarian hyperstimulation syndrome: a novel approach. Reprod Biomed Online. 2006 Aug;13(2):194-7. doi: 10.1016/s1472-6483(10)60614-1. PMID 16895631
- [Background] Hostalek U, Campbell I. Metformin for diabetes prevention: update of the evidence base. Curr Med Res Opin. 2021 Oct;37(10):1705-1717. doi: 10.1080/03007995.2021.1955667. Epub 2021 Jul 28. PMID 34281467
- [Background] Praharaj SK, Jana AK, Goyal N, Sinha VK. Metformin for olanzapine-induced weight gain: a systematic review and meta-analysis. Br J Clin Pharmacol. 2011 Mar;71(3):377-82. doi: 10.1111/j.1365-2125.2010.03783.x. PMID 21284696
- [Background] Sivalingam VN, Myers J, Nicholas S, Balen AH, Crosbie EJ. Metformin in reproductive health, pregnancy and gynaecological cancer: established and emerging indications. Hum Reprod Update. 2014 Nov-Dec;20(6):853-68. doi: 10.1093/humupd/dmu037. Epub 2014 Jul 10. PMID 25013215
- [Background] Arslanian S, Bacha F, Grey M, Marcus MD, White NH, Zeitler P. Evaluation and Management of Youth-Onset Type 2 Diabetes: A Position Statement by the American Diabetes Association. Diabetes Care. 2018 Dec;41(12):2648-2668. doi: 10.2337/dci18-0052. No abstract available. PMID 30425094
- [Background] Yari S, Khoei HH, Saber M, Esfandiari F, Moini A, Shahhoseini M. Metformin attenuates expression of angiogenic and inflammatory genes in human endometriotic stromal cells. Exp Cell Res. 2021 Jul 15;404(2):112659. doi: 10.1016/j.yexcr.2021.112659. Epub 2021 May 19. PMID 34022204
- [Background] Stochino-Loi E, Major AL, Gillon TER, Ayoubi JM, Feki A, Bouquet de Joliniere J. Metformin, the Rise of a New Medical Therapy for Endometriosis? A Systematic Review of the Literature. Front Med (Lausanne). 2021 May 11;8:581311. doi: 10.3389/fmed.2021.581311. eCollection 2021. PMID 34046415
- [Background] Kimber-Trojnar Z, Dluski DF, Wierzchowska-Opoka M, Ruszala M, Leszczynska-Gorzelak B. Metformin as a Potential Treatment Option for Endometriosis. Cancers (Basel). 2022 Jan 24;14(3):577. doi: 10.3390/cancers14030577. PMID 35158846
- [Background] Hopkins BD, Goncalves MD, Cantley LC. Insulin-PI3K signalling: an evolutionarily insulated metabolic driver of cancer. Nat Rev Endocrinol. 2020 May;16(5):276-283. doi: 10.1038/s41574-020-0329-9. Epub 2020 Mar 3. PMID 32127696
- [Background] Dinulescu DM, Ince TA, Quade BJ, Shafer SA, Crowley D, Jacks T. Role of K-ras and Pten in the development of mouse models of endometriosis and endometrioid ovarian cancer. Nat Med. 2005 Jan;11(1):63-70. doi: 10.1038/nm1173. Epub 2004 Dec 26. PMID 15619626
- [Background] Anglesio MS, Papadopoulos N, Ayhan A, Nazeran TM, Noe M, Horlings HM, Lum A, Jones S, Senz J, Seckin T, Ho J, Wu RC, Lac V, Ogawa H, Tessier-Cloutier B, Alhassan R, Wang A, Wang Y, Cohen JD, Wong F, Hasanovic A, Orr N, Zhang M, Popoli M, McMahon W, Wood LD, Mattox A, Allaire C, Segars J, Williams C, Tomasetti C, Boyd N, Kinzler KW, Gilks CB, Diaz L, Wang TL, Vogelstein B, Yong PJ, Huntsman DG, Shih IM. Cancer-Associated Mutations in Endometriosis without Cancer. N Engl J Med. 2017 May 11;376(19):1835-1848. doi: 10.1056/NEJMoa1614814. PMID 28489996
- [Background] Becker CM, Gattrell WT, Gude K, Singh SS. Reevaluating response and failure of medical treatment of endometriosis: a systematic review. Fertil Steril. 2017 Jul;108(1):125-136. doi: 10.1016/j.fertnstert.2017.05.004. PMID 28668150
- [Background] Olive DL. Medical therapy of endometriosis. Semin Reprod Med. 2003 May;21(2):209-22. doi: 10.1055/s-2003-41327. PMID 12917790
- [Background] Shim JY, Laufer MR. Adolescent Endometriosis: An Update. J Pediatr Adolesc Gynecol. 2020 Apr;33(2):112-119. doi: 10.1016/j.jpag.2019.11.011. Epub 2019 Dec 5. PMID 31812704
- [Background] Hoshiai H, Ishikawa M, Sawatari Y, Noda K, Fukaya T. Laparoscopic evaluation of the onset and progression of endometriosis. Am J Obstet Gynecol. 1993 Sep;169(3):714-9. doi: 10.1016/0002-9378(93)90649-4. PMID 8372885
- [Background] DiVasta AD, Vitonis AF, Laufer MR, Missmer SA. Spectrum of symptoms in women diagnosed with endometriosis during adolescence vs adulthood. Am J Obstet Gynecol. 2018 Mar;218(3):324.e1-324.e11. doi: 10.1016/j.ajog.2017.12.007. Epub 2017 Dec 13. PMID 29247637
- [Background] Pugsley Z, Ballard K. Management of endometriosis in general practice: the pathway to diagnosis. Br J Gen Pract. 2007 Jun;57(539):470-6. PMID 17550672
- [Background] Ballweg ML. Big picture of endometriosis helps provide guidance on approach to teens: comparative historical data show endo starting younger, is more severe. J Pediatr Adolesc Gynecol. 2003 Jun;16(3 Suppl):S21-6. doi: 10.1016/s1083-3188(03)00063-9. No abstract available. PMID 12742183
- [Background] Simoens S, Hummelshoj L, D'Hooghe T. Endometriosis: cost estimates and methodological perspective. Hum Reprod Update. 2007 Jul-Aug;13(4):395-404. doi: 10.1093/humupd/dmm010. PMID 17584822
- [Background] Soliman AM, Surrey E, Bonafede M, Nelson JK, Castelli-Haley J. Real-World Evaluation of Direct and Indirect Economic Burden Among Endometriosis Patients in the United States. Adv Ther. 2018 Mar;35(3):408-423. doi: 10.1007/s12325-018-0667-3. Epub 2018 Feb 15. PMID 29450864
- [Background] Bulletti C, Coccia ME, Battistoni S, Borini A. Endometriosis and infertility. J Assist Reprod Genet. 2010 Aug;27(8):441-7. doi: 10.1007/s10815-010-9436-1. Epub 2010 Jun 25. PMID 20574791
- [Background] Shafrir AL, Farland LV, Shah DK, Harris HR, Kvaskoff M, Zondervan K, Missmer SA. Risk for and consequences of endometriosis: A critical epidemiologic review. Best Pract Res Clin Obstet Gynaecol. 2018 Aug;51:1-15. doi: 10.1016/j.bpobgyn.2018.06.001. Epub 2018 Jul 3. PMID 30017581